CLINICAL TRIAL: NCT04089592
Title: Comparison Of Dexmedetomidine and Fentanyl In Attenuation Of Hemodynamic Response To Direct Laryngoscopy And Intubation In Patient Undergoing Laparoscopic Cholecystectomy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Sana Urooj, Assistant Professor, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SUrooj
Record Dates: First submitted 2019-08-22; First posted 2019-09-13 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Cholecystectomy; Elective Surgery
Keywords: Laparoscopic Cholecystectomy; Dexmedetomidine; Fentanyl; Hemodynamics response; Direct laryngoscopy; Intubation
MeSH Terms: interventions — Dexmedetomidine; Fentanyl

STUDY DESIGN:
Intervention Model Description: RCT, Double-blind, Randomized control trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patient meeting the inclusion criteria will be randomly allocated divided into two groups by chit paper method A, B (30 participants in each group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dex Group (Experimental): intravenous dexmedetomidine 0.6mcg/kg in 100ml normal saline 0.9%
  Interventions: Drug: Dexmedetomidine
- Fent Group (Experimental): intravenous fentanyl at 2mcg/kg in 100ml saline
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Dexmedetomidine — intravenous dexmedetomidine 0.6mcg/kg in 100ml normal saline 0.9%
  Other Names: Fentanyl
  Arms: Dex Group
Drug: Fentanyl — intravenous fentanyl at 2mcg/kg in 100ml saline
  Other Names: Dexmedetomidine
  Arms: Fent Group

SUMMARY:
Compare effects of intravenous dexmedetomidine and fentanyl in attenuation of intubation response in a patient undergoing laparoscopic cholecystectomy.

Compare the effects of intravenous dexmedetomidine and fentanyl in sedation, perioperative complications, and recovery in these patients.

Dexmedetomidine is comparatively a newer drug in countries like Pakistan. There is no research work available at the national level and scarcity of data at an international level with inconclusive outcomes. Our participation in the form of this research will add to scientific literature and step up ahead at the international level.

Fentanyl citrate is a narcotic analgesic interacting predominantly with the opioid μ receptor and exerting its principal pharmacological effect on CNS. Its primary action of therapeutic value is analgesia and sedation. It is extensively used for anesthetic and analgesic most often in operating room and ICU.

DETAILED DESCRIPTION:
This is double-blind, a single centered randomized clinical trial which is based on assessing the hemodynamic stability provided by our study drugs during laryngoscopy and intubation in a patient undergoing laparoscopic cholecystectomy. In addition to that this study will assess the perioperative complication and postoperative recovery in these patients. Laparoscopy has now become the standard technique of choice for cholecystectomy which results in pathophysiological changes characterized by an increase in arterial pressure and heart rate (HR). Many types of research have been done in an attempt to minimize adverse effects by adding adjuvants to the conventional method of general anesthesia. Our research is also based on this aim. The objective of this study to determine the hemodynamic stability during laryngoscopy and intubation, peri-operative complication and post-operative recovery. The patients will be divided into two groups randomly and will be given the desired drugs via intravenous line by on floor consultant anesthetist who will be blinded to the drug. The study subjects' hemodynamics will be observed until 10 minutes of intubation. Any perioperative complication will be noted. The subjects will also be followed postoperatively in recovery to check there sedation score and recovery (Aldrete score) will be noted after 10 minutes after the patient shifted to recovery.

ELIGIBILITY:
Inclusion Criteria:

1. ASA-I and ll patients
2. Male and female patient of age 20-70 years.
3. Undergoing Elective laparoscopic cholecystectomy.

Exclusion Criteria:

1. Pregnant and lactating females
2. Short thick neck with anticipated difficult intubation.
3. Obese patients.
4. Narcotic addicts.
5. Full stomach patient or with higher chances of aspiration.
6. Patient allergic to any of the study medications.
7. Patients high risk to develop serotonin syndrome. (patient taking an antidepressant and other psychomotor medications.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | at Baseline
  Hemodynamic response(induction) will be assessed on different point in time during procedure
Systolic blood pressure | 0 minute
  Hemodynamic response(induction) will be assessed on different point in time during procedure
Systolic blood pressure | 1 minute
  Hemodynamic response(induction) will be assessed on different point in time during procedure
Systolic blood pressure | 3 minute
  Hemodynamic response(induction) will be assessed on different point in time during procedure
Systolic blood pressure | 5 minute
  Hemodynamic response(induction) will be assessed on different point in time during procedure
Systolic blood pressure | 10 minute
  Hemodynamic response(induction) will be assessed on different point in time during procedure
Diastolic blood pressure | at Baseline
  Hemodynamic response(induction) will be assessed on different point in time during procedure
Diastolic blood pressure | 0 minute
  Hemodynamic response(induction) will be assessed on different point in time during procedure
Diastolic blood pressure | at 1 minute
  Hemodynamic response(induction) will be assessed on different point in time during procedure
Diastolic blood pressure | at 3 minutes
  Hemodynamic response(induction) will be assessed on different point in time during procedure
Diastolic blood pressure | at 5 minutes
  Hemodynamic response(induction) will be assessed on different point in time during procedure
Diastolic blood pressure | at 10 minutes
  Hemodynamic response(induction) will be assessed on different point in time during procedure
Heart rate | at Baseline
  Hemodynamic response(induction) will be assessed on different point in time during procedure
Heart rate | at 0 minute
  Hemodynamic response(induction) will be assessed on different point in time during procedure
Heart rate | at 1 minute
  Hemodynamic response(induction) will be assessed on different point in time during procedure
Heart rate | at 3 minutes
  Hemodynamic response(induction) will be assessed on different point in time during procedure
Heart rate | 5 minutes
  Hemodynamic response(induction) will be assessed on different point in time during procedure
Heart rate | at 10 minutes
  Hemodynamic response(induction) will be assessed on different point in time during procedure
Mean atrial pressure | at Baseline
  Hemodynamic response(induction) will be assessed on different point in time during procedure
Mean atrial pressure | at 0 minute
  Hemodynamic response(induction) will be assessed on different point in time during procedure
Mean atrial pressure | at 1 minute
  Hemodynamic response(induction) will be assessed on different point in time during procedure
Mean atrial pressure | at 3 minute
  Hemodynamic response(induction) will be assessed on different point in time during procedure
Mean atrial pressure | at 5 minute
  Hemodynamic response(induction) will be assessed on different point in time during procedure
Mean atrial pressure | at 10 minute
  Hemodynamic response(induction) will be assessed on different point in time during procedure
SpO (oxygen saturation) | at Baseline
  Hemodynamic response(induction) will be assessed on different point in time during procedure
SpO (oxygen saturation) | at 0 minute
  Hemodynamic response(induction) will be assessed on different point in time during procedure
SpO (oxygen saturation) | at 1 minute
  Hemodynamic response(induction) will be assessed on different point in time during procedure
SpO (oxygen saturation) | at 3 minute
  Hemodynamic response(induction) will be assessed on different point in time during procedure
SpO (oxygen saturation) | at 5 minute
  Hemodynamic response(induction) will be assessed on different point in time during procedure
SpO (oxygen saturation) | at 10 minute
  Hemodynamic response(induction) will be assessed on different point in time during procedure

SECONDARY OUTCOMES:
Ramsey score | at arrival
  Sedation scale with minimum score 1 indicate good response and maximum score 6 worst response
Ramsey score | at 10 minutes
  Sedation scale with minimum score 1 indicate good response and maximum score 6 worst response
Aldrete score | at arrival
  Post anesthesia Recovery assessment scale with minimum score 0 indicate worst response and maximum score 10 indicate excellent recovery
Aldrete score | at 10 min
  Post anesthesia Recovery assessment scale with minimum score 0 indicate worst response and maximum score 10 indicate excellent recovery
Complications | Will be assessed within Hospital stay at follow for 1 week
  Post operative complication
Laryngospasm | Will be assessed within Hospital stay at follow for 1 week
  Post operative complication
Bradycardia | Will be assessed within Hospital stay at follow for 1 week
  Post operative complication
Regurgitation | Will be assessed within Hospital stay at follow for 1 week
  Post operative complication
Post operative vomiting and nausea | Will be assessed within Hospital stay at follow for 1 week
  Post operative complication
Hypertension | Will be assessed within Hospital stay at follow for 1 week
  Post operative complication
Hypotension | Will be assessed within Hospital stay at follow for 1 week
  Post operative complication

CONTACTS AND LOCATIONS:
Overall Officials: Sana Urooj, FCPS, Principal Investigator — Dr. Ruth K.M. Pfau Civil Hospital, Karachi
Locations (2):
- Pakistan (2):
  - Civil Hospital Karachi, Karachi, Sindh
  - DUHS, Civil hospital Karachi (CHK), Karachi, Sindh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vaswani JP, Debata D, Vyas V, Pattil S. Comparative Study of the Effect of Dexmedetomidine Vs. Fentanyl on Haemodynamic Response in Patients Undergoing Elective Laparoscopic Surgery. J Clin Diagn Res. 2017 Sep;11(9):UC04-UC08. doi: 10.7860/JCDR/2017/27020.10578. Epub 2017 Sep 1. PMID 29207810